CLINICAL TRIAL: NCT04760964
Title: Mitochondrial DAMPs as Mechanistic Biomarkers of Mucosal Inflammation in Crohn's Disease and Ulcerative Colitis (MUSIC)
Brief Title: Mitochondrial DAMPs as Mechanistic Biomarkers of Mucosal Inflammation in Crohn's Disease and Ulcerative Colitis
Acronym: MUSIC
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC19037
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — SALIVA: 1 sample for DNA sampling. BLOOD: At each time point, ~40mls of blood will be taken. Serum for normal IBD care and Mediators/Biomarkers, Serum proteins and LC-MS EDTA tubes for normal IBD care and Mediators/metabolites/biomarkers RNA tube (PAXgene®) for RNA sequencing of host transcriptome ILEO-COLONOSCOPY SAMPLES: Standard research sampling involves: 4 biopsies (2 for formalin fixation and 2 for RNA-later) from ileum (the small bowel), caecum, transverse colon and rectum respectively. Total of 16 biopsies.
  STOOL SAMPLES: For Microbiome Next Generation Sequencing/Calprotectin/Stool biomarkers and faecal immunochemical test (FIT)
  In selected patients:
  BLOOD SAMPLES: 10-20 participants with anticipated high DAMP release. ~10-20 IBD patients with inactive, quiescent disease.
  SURGICAL SAMPLES: Surplus tissue may be obtained from specimens of the colon and ileum that have been surgically removed either at the time of operation or during histopathological evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MUSIC study is a multi-centre, longitudinal study set in the real world IBD clinical setting to investigate and develop a new biomarker approach that aims to inform both patients and clinicians of the current state of the affected gut lining (how inflamed or whether the bowel wall has completely healed).

This new biomarker approach will study a panel of molecular signs in IBD patients' blood, stools and biopsies that will be correlated to the current gold standard of direct gut visual examination using ileo-colonoscopy and flexible sigmoidoscopy tests (a fibre-optic examination of the lower small bowel and large bowel). Here, the state and appearances of IBD patients' gut lining will be assessed over one year in response to treatment given to them by their NHS IBD consultant.

This approach will focus on the role of damage associated molecular patterns (DAMPs), also known as 'danger signals'. DAMPs are found in our own cells and are released during tissue stress or injury. Like signals from bacteria, they can trigger inflammation. In the MUSIC study, blood, stool, saliva and gut samples obtained from participants during active IBD and in clinical remission will be used in order to understand how DAMPs contribute to the development of gut inflammation.

DETAILED DESCRIPTION:
The hypothesis is that mitochondrial DAMPs are good mechanistic biomarkers for mucosal inflammation and healing in IBD.

Complete mucosal healing (total resolution and absence of ulcerations in the gut) is the most sought-after treatment target with the best long-term implication in prognosis.

Up to now IBD clinicians rely on (1) clinical symptoms (how patients feel, their bowel habit, presence of blood in stools), (2) clinical tests such as stool calprotectin (FC) and blood C-reactive protein (CRP) to inform both themselves and the patients, how well the drug treatment is working and importantly, whether the ulcers and inflammation seen in the gut lining have healed or not.

Current evidence shows that these approaches are not fully informative. For example, 30% of patients with significant subjective improvement in their symptoms following treatment of active CD have evidence of active inflammation in their gut lining when further assessed with an ileo-colonoscopy. Blood and stool tests to predict mucosal healing are only useful in around 60-70% and very limited, in guiding the doctors in how severely inflamed the bowel wall is during active IBD.

Direct visualisation using ileo-colonoscopy or flexible sigmoidoscopy is the most accurate approach to assess disease activity and mucosal healing in response to medical treatment. By knowing precisely, how the gut wall inflammation is responding to treatment, the clinician can accurately manage the IBD patient (by either changing the dose and type of treatment, and whether to carry on with expensive, strong medications with potentially serious side effects). However, in the real world, follow-up endoscopic tests are difficult to carry out as they are expensive and we lack the capacity to undertake these examinations within NHS.

Project Goals

The main goal for the MUSIC study is to investigate the role of mitochondrial DAMPs in the clinic as an indicator of gut inflammation and subsequent mucosal healing in response to medical treatment in IBD.

Secondly, further scientific studies will be carried out using blood, stool, saliva and gut biopsy samples to investigate how mitochondrial DAMPs (and all known biomarkers and biological data such as genetics) contribute to the abnormal development of gut inflammation in IBD.

Primary research questions:

* Do mitochondrial DAMPs predict the activity and severity of IBD-inflammation?
* Does normalisation of mitochondrial DAMPs reflect complete endoscopic mucosal healing in IBD?
* How do mitochondrial DAMPs compare to current biomarkers (FC, CRP) and clinical symptoms (HBI/Mayo Score) in assessing IBD inflammation and mucosal healing?
* Can a simple decision-making model be developed to predict mucosal healing based on mitochondrial DAMPs, together with relevant biological data such as genetics, blood transcriptomics, microbiome; and current clinical biomarkers such as calprotectin, faecal haemoglobin and blood CRP?

Secondary research questions:

* How are mitochondrial DAMPs released from cells in the IBD gut?
* What types of cells are important in mitochondrial DAMP release? There are many forms of inflammatory cells in affected IBD gut (e.g. macrophage, epithelial, neutrophils). It is possible that different cell types may contain more inflammatory DAMPs.
* Which type of mitochondrial DAMPs are important in causing inflammation? Can mitochondrial DAMPs pinpoint a specific underlying genetic susceptibility (e.g. autophagy) or inflammatory mechanism in IBD?

Rationale

The focus is to investigate mitochondrial DAMPs' utility in two clinically relevant scenarios: (a) How severe or active is the disease? (b) How well are we treating IBD? - with endoscopic endpoints of mucosal inflammation and healing respectively. The Simple Endoscopic Score for Crohn's Disease (SES-CD) and Endoscopic Mayo Score (eMS) will be used for CD and UC respectively. Both have been validated and used widely in research and in clinical trials. By using these objective endoscopic endpoints, mtDAMPs (and in combination with current biomarkers FC and CRP) can be tested across a range of mucosal inflammation (full healing to severe).

In addition to this, it will be investigated if mitochondrial DAMPs can identify a subclinical pathogenic mechanism (e.g. [a] defective autophagy to clear damaged mitochondria; [b] de-regulated innate immune response to mitochondrial DAMPs.) These data will pave the way for future use of mitochondrial DAMP biomarkers as part of a stratified approach for new treatments targeted at mitochondrial DAMPs and their downstream inflammatory mechanisms in IBD.

Study Population

Presently within usual NHS care, all patients with active IBD, especially those to be initiated on biologic or immunomodulator treatment, are followed up where they will have documentation of disease activity (Harvey Bradshaw Index [HBI] or UC Mayo Score [MS], stool calprotectin, C-reactive protein, albumin and blood count) to assess their well-being and response to medical treatment.

With MUSIC, patients will be followed up prospectively (aligning the usual NHS clinical care above) and will receive additional endoscopic follow-up to assess mucosal healing in response to medical treatment. Thus, the MUSIC study will incorporate a prospective endoscopic evaluation of mucosal inflammation and mucosal healing into IBD clinics.

The recruitment and subsequent clinical data and sample collection will take place at 0, 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be able to give consent and aged 16 years old and over.
2. All patients must have a diagnosis of IBD (CD or UC)
3. All patients must have active IBD at the time of screening:

   • Active IBD symptoms by referring clinician's judgement in addition to one of the below criteria (within 6 weeks of screening):
   * FC level of >100ug/g
   * Blood CRP >5mg/l
   * Endoscopic, radiological or histological evidence of active IBD
4. All IBD patients with disease involvement that is amenable for endoscopic assessment of mucosal healing. This includes:

   * CD patients with previous ileal or colonic surgical resection
   * CD patients with perianal disease where ileo-colonoscopy or sigmoidoscopy are not contraindicated
   * CD patients with ileal involvement only where endoscopic disease activity can be recorded
5. All IBD patients will require a recent ileo-colonoscopy or flexible sigmoidoscopy within 6 weeks of recruitment that has:

   * Clear documentation of endoscopic disease activity and extent (SES-CD and Rutgeert's score for CD; Mayo Score or UCEIS for UC)
   * Photographs of endoscopic mucosal IBD disease activity
   * If there is not a recent ileo-colonoscopy or flexible sigmoidoscopy, the participant will be asked to undergo an ileo-colonoscopy or flexible sigmoidoscopy at baseline.
6. If patients have undergone an ileo-colonoscopy or flexible sigmoidoscopy within 6 weeks but with an endoscopic report that is insufficient in endoscopic disease activity data as per (5), potential participant can still be considered providing there is:

   * Supporting objective evidence of IBD disease activity (FC, CRP) within 2 weeks of index ileo-colonoscopy or flexible sigmoidoscopy.

Exclusion Criteria:

1. IBD patients with severe/fulminant disease at screening:

   * Subjects with colitis fulfilling the Truelove and Witts' criteria (stool frequency >6/24 hours with all of the features of fever >38C, pulse rate >100 beats per minute, blood haemoglobin <105 g/l, albumin <30g/l)
   * Subjects displaying evidence of toxic megacolon (transverse colon diameter >6m on plain abdominal X-ray with accompanying full radiological report). Note - abdominal X-ray will be carried out if clinically indicated by referring clinician
   * Evidence of significant bowel obstruction, abdominal sepsis, abscess formation and fistula formation (bowel or perianal) as documented by referring clinician that is supported by clinical, radiological and blood laboratory investigations
2. Referring clinician's judgement where surgical intervention (colectomy or resection) is deemed likely within 3 months of screening
3. Evidence of intestinal dyplasia or malignancy (histologic, endoscopic or radiologic)
4. UC patients with limited involvement of the rectum (<15cm - proctitis)
5. UC patients who have had a colectomy (total and subtotal)
6. UC patients with an ileo-anal pouch
7. IBD (UC, CD or IBD-U) with an intestinal stoma
8. Patients where ileo-colonoscopy or flexible sigmoidoscopy are contra-indicated (e.g. significant co-morbidities e.g. cardiovascular, respiratory, cancer, renal failure; and pregnancy)
9. Participants where there are limitations to language communication where there is a potential issue where information sheet cannot be reliably understood and/or the subject cannot provide full informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants will have active IBD at the time of recruitment.
  The aim is to capture a wide spectrum of IBD patients with active disease, hence strict criteria for IBD disease severity/extent/activity is not applied.
  However, suitable potential participants must have active IBD based on clinical evaluation of referring clinician and any one of the below from investigations which have been carried out within 6 weeks of screening:
  1. FC level of >100ug/g
  2. Blood CRP >5mg/l
  3. Endoscopic, radiological or histological evidence of active IBD
  There will be 2 main groups:
  1. IBD patients with acute flare requiring medical treatment (corticosteroids, immunomodulator or biologics)
  2. IBD patients on established medical treatments (biologics or immunomodulators) that require a change due to poor control of disease activity
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The role of mitochondrial DAMPs as an indicator of gut inflammation and mucosal healing | 12 months
  To investigate the role of mitochondrial DAMPs in the clinic as an indicator of gut inflammation and subsequent mucosal healing in response to medical treatment in IBD.

CONTACTS AND LOCATIONS:
Overall Officials: Gwo-Tzer Ho, Principal Investigator — University of Edinburgh
Locations (3):
- United Kingdom (3):
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - NHS Greater Glasgow & Clyde, Glasgow

IPD SHARING:
Plan to Share IPD: Undecided